CLINICAL TRIAL: NCT01396369
Title: Impact of Flaxseed Lignan (Brevail) on Polycystic Ovarian Syndrome
Brief Title: Flaxseed Lignan (Brevail)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12459
Record Dates: First submitted 2011-07-14; First posted 2011-07-18 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Polycystic Ovarian Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Birth control (Active Comparator)
  Interventions: Drug: Birth control
- Birth control plus Brevail (Experimental)
  Interventions: Drug: Birth control plus Brevail

INTERVENTIONS:
Drug: Birth control — In the initial visit, History and Physical Exam,menstrual history, pregnancy history, documentation of hirsutism using Ferriman-Gallwey scoring,body weight, height, and body mass index.The baseline ultrasound blood tests. After the lab tests, the patients in the control group will be started on OC (standard clinical practice) and those in the treatment group will be started on OC with Brevail (2 pills once a day). The patients will return to the clinic for a follow up visit after 3 months. If no side effects, Brevail and OC will be continued for 3 more months. The control group will also have a follow up after 3 months of OC. Six months after the initiation of the study, the patients in the both groups will have another H&P as well as repeat ultrasound and blood tests.
  Arms: Birth control
Drug: Birth control plus Brevail — In the initial visit, History and Physical Exam,menstrual history, pregnancy history, documentation of hirsutism using Ferriman-Gallwey scoring,body weight, height, and body mass index.The baseline ultrasound blood tests. After the lab tests, the patients in the control group will be started on OC (standard clinical practice) and those in the treatment group will be started on OC with Brevail (2 pills once a day). The patients will return to the clinic for a follow up visit after 3 months. If no side effects, Brevail and OC will be continued for 3 more months. The control group will also have a follow up after 3 months of OC. Six months after the initiation of the study, the patients in the both groups will have another H&P as well as repeat ultrasound and blood tests.
  Arms: Birth control plus Brevail

SUMMARY:
PCOS is a disorder which is characterized by hyperandrogenism (high serum male hormone levels), ovulatory dysfunction, and polycystic ovaries (multiple follicles-over 12- in the ovary). There is no universally accepted definition for PCOS. The Rotterdam criteria require 2 of 3 criteria for diagnosis, including hyperandrogenism (clinical hirsutism or serum hormone measurement), oligomenorrhea/amenorrhea, and ultrasound findings of polycystic ovaries.

This study is a prospective randomized pilot study designed to evaluate the effects of flaxseed supplementation (with Brevail) on hormonal and lipid metabolism balance in polycystic ovarian syndrome (PCOS) patients.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 to 40 year old female with:
* Diagnosis of PCOS by menstrual irregularity (fewer than 9 menses annually/interval over 40 days), Ferriman-Galleway score >8, and/or hyperandrogenemia defined as total testosterone >80ng/dl or bioavailable testosterone >8.4 ng/dl.
* Mentally competent.

Exclusion Criteria:

* Use of oral contraceptives, spironolactone, or insulin-sensitizing agents within the past 2 months.
* Long-term or chronic use of oral antibiotics.
* Hysterectomy.
* FSH >15.
* Pregnancy/lactation.
* Consumption of flaxseed within the last month.
* Diagnosis of thyroid disease, nonclassical adrenal hyperplasia, and hyperprolactinemia.
* Use of any dietary fiber supplements which are newly started (within the past 6 months) and agreement not to use any new fiber supplements during the study period.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2011-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Primary outcomes to assess are the changes of testosterone levels and hirsutism. | up to 6 months

SECONDARY OUTCOMES:
Secondary outcomes to assess are the lipid profile and estrogen levels. | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sam Kim, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States